CLINICAL TRIAL: NCT02226354
Title: Study of the Safety and Efficacy of Dietary Buglossoides Oil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Réseau de Santé Vitalité Health Network (Other)
Responsible Party: Principal Investigator, Marc Surette, Professor, Réseau de Santé Vitalité Health Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HC-NHPD-196699
Record Dates: First submitted 2014-08-06; First posted 2014-08-27 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Dietary vegetable oil; Stearidonic acid; Tissue; Fatty Acid; composition
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flaxseed oil (Active Comparator): 9.73ml Flaxseed oil once daily, for 28 days
  Interventions: Dietary Supplement: Flaxseed oil
- Ahiflower oil (Experimental): 9.73ml Ahiflower oil once daily, for 28 days
  Interventions: Dietary Supplement: Ahiflower oil

INTERVENTIONS:
Dietary Supplement: Ahiflower oil — 9.73 ml per day for 28 days
  Other Names: Buglossoides oil; Buglossoides arvensis oil
  Arms: Ahiflower oil
Dietary Supplement: Flaxseed oil — 9.73ml per day for 28 days
  Other Names: Linseed oil
  Arms: Flaxseed oil

SUMMARY:
Seeds from the Buglossoides arvensis plant (trademarked as Ahiflower™) produce oil that is a rich natural source (20%) of stearidonic acid (SDA), a metabolic intermediate between omega-3 fatty acids found in other plants (such as flax) and those found in fish oils.

The objectives of this study to collect safety data and to investigate the accumulation of long chain n-3 polyunsaturated fatty acids in human lipids following oral supplementation with Ahiflower oil in healthy adults.

DETAILED DESCRIPTION:
This is a single-center, randomized, comparator-controlled, double-blind study in healthy subjects. Forty subjects will be randomly assigned to 2 supplementation groups (n=20 per group). One group will consume 10 ml of Buglossoides oil daily and one group will consume 10 ml of flax seed oil daily for a 4 week period. Baseline data will be obtained at week 0. Subjects will return to the clinic after 2 weeks and again after 4 weeks for measurement of safety and efficacy endpoints.

The efficacy parameters are statistically significant changes from baseline and between groups in plasma, red blood cell and leukocyte omega-3 fatty acid content.

The primary efficacy endpoint will be:

Plasma EPA concentration expressed as μmol/L plasma.

The secondary efficacy endpoints will be:

1. Plasma 20:4n-3 and DPA individually as μmol/L;
2. Plasma 20:4n-3, EPA and DPA individually as % of total fatty acids;
3. Erythrocyte 20:4n-3, EPA and DPA individually as % of total fatty acids;
4. Mononuclear cell 20:4n-3, EPA and DPA individually as % of total fatty acids;
5. Neutrophil 20:4n-3, EPA and DPA individually as % of total fatty acids;
6. The omega-3 index (defined as the sum of red blood cell EPA and DHA concentrations), expressed as % total fatty acids.

Safety endpoints will be:

1. fasting serum chemistry
2. fasting hematology profile
3. fasting blood lipid profile

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women, using an effective form of birth control (such as oral contraceptives, injectable contraceptives or the barrier method such as a intrauterine device (IUD) with a spermicide, a diaphragm with a spermicide, a condom with a spermicide or a sponge with a spermicide) for at least 3 months prior to entry into the study and continuing during participation in the study.
* 18 to 65 years of age, inclusive.
* Body mass index (BMI) 18 - 35 kg/m2
* Subject is willing to avoid alcohol consumption for 24h prior to every clinic visit.
* The subject will not modify smoking habits during supplementation period.
* No significant medical conditions that in the opinion of the qualified physician, would preclude the subject's participation in the study.
* Signed informed consent.
* Willing to follow all study procedures including study visits, fasting blood draws, stable body weight, normal eating habits, current activity level, and compliance with study preparation.
* Willing to not consume fish, crustaceans and shellfish for the duration of the study.

Exclusion Criteria:

* Pregnancy or lactation. Women trying to conceive. Women who will try to conceive who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. Method of contraception must be recorded in the case report file.
* Individual has a condition the study physician believes would interfere with the participant's ability to provide informed consent, comply with his responsibilities during the study, which might confound the interpretation of the study results or put the person at undue risk.
* Medical conditions including an active peptic ulcer, inflammatory bowel disease, or gastrointestinal bleeding and any medical condition or prior gastrointestinal surgery that could influence absorption, metabolism or excretion of the study supplement.
* History or presence of significant, renal, hepatic, gastrointestinal, pulmonary, biliary, neurological or endocrine disorders.
* History or presence of cancer in the past 2 yrs, except for non-melanoma skin cancers (e.g. basal or squamous cell carcinoma of the skin).
* Clinically significant abnormal laboratory test results including but not limited to LDL-cholesterol ≥ 4.1mM, triglyceride levels ≥3.95mM, fasting creatinine ≥ 1.5 mg/dL, alkaline phosphatase or aspartate aminotransferase ≥ 1.5 times the upper limit of normal.
* Currently being treated for angina, arrhythmia and/or congestive heart failure. History of myocardial infarction or stroke.
* Presence of coronary heart disease or presence of multiple risk factors that result in a greater than 20% chance for developing coronary artery disease within 10 years using the Framingham risk index.
* Uncontrolled hypertension (resting systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
* Type 1 or 2 diabetes. Fasting glucose ≥ 100 mg/dL. HbA1c ≥ 6.0.
* If a smoker, subject smokes no more than 1 pack (20 cigarettes) daily.
* History (within 12 months) or current alcohol or substance abuse (no more than 14 consumptions per week; 1 consumption= 12 oz beer, 5 oz wine, 1.5 oz distilled spirits).
* Use of any lipid-altering medications (statins, bile acid sequestrants, cholesterol absorption inhibitors, fibrates, prescription formulations of niacin).
* Unstable use of thyroid medication. Stable, treated hypothyroidism is not an exclusion criteria.
* Use of any weight loss or lipid metabolism medication/supplement/program (including lipase inhibitors) within 1 month of study period OR weight gain or loss > 2 kg in the past 3 months.
* Currently taking fish oil or any other omega-3 or omega-6 polyunsaturated fatty acid supplement/drug within three months of Visit 1 and throughout the study. Consumption of fatty fish (salmon, herring, mackerel, albacore tuna, and sardines) more than twice a month within three months of visit 1 and throughout the study period. Consumption (more than twice a month) of any EPA/DHA enriched foods (e.g. DHA-enriched eggs) within three months of Visit 1. Unwillingness to avoid all fish including shellfish and crustaceans throughout the study period.
* Use of alpha-linolenic acid-containing seeds and oils such as flax seed, perilla seed, hemp, spirulina, walnut, mustard seed or black currant seeds/oil within three months of Visit 1 and throughout the study.
* Use of an investigational product within the previous 30 days.
* Has donated blood up to 8 weeks before the start of the study. Not willing to cease being a blood donor during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Plasma eicosapentaenoic acid (EPA) concentration | Day 0, Day 14, Day 28
  Expressed as μmol/L plasma

SECONDARY OUTCOMES:
Plasma eicosatetraenoic acid (ETA) concentration | Day 0, Day 14, Day 28
  Expressed as μmol/L
Plasma docosapentaenoic acid (DPA) concentration | Day 0, Day 14, Day 28
  Expressed as μmol/L
Plasma 20:4n-3, EPA and DPA individually as % of total fatty acids | Day 0, Day 14, Day 28
Erythrocyte 20:4n-3, EPA and DPA individually as % of total fatty acids | Day 0, Day 14, Day 28
Mononuclear cell 20:4n-3, EPA and DPA individually as % of total fatty acids | Day 0, Day 14, Day 28
Neutrophil 20:4n-3, EPA and DPA individually as % of total fatty acids | Day 0, Day 14, Day 28
Omega-3 index (defined as the sum of red blood cell EPA and DHA concentrations) | Day 0, Day 14, Day 28
  Expressed as % total fatty acids
Fasting serum chemistry: glucose | Day 0, Day 14, Day 28
Fasting serum chemistry: calcium | Day 0, Day 14, Day 28
Fasting serum chemistry: sodium | Day 0, Day 14, Day 28
Fasting serum chemistry: potassium | Day 0, Day 14, Day 28
Fasting serum chemistry: blood urea nitrogen | Day 0, Day 14, Day 28
Fasting serum chemistry: creatinine | Day 0, Day 14, Day 28
Fasting serum chemistry: alkaline phosphatase | Day 0, Day 14, Day 28
Fasting serum chemistry: aspartate aminotransferase | Day 0, Day 14, Day 28
Fasting serum chemistry: gamma-glutamyl transferase | Day 0, Day 14, Day 28
Fasting serum chemistry: total bilirubin | Day 0, Day 14, Day 28
Fasting serum chemistry: amylase | Day 0, Day 14, Day 28
Fasting serum chemistry: uric acid | Day 0, Day 14, Day 28
Fasting serum chemistry: albumin | Day 0, Day 14, Day 28
Fasting hematology profile: white blood cell count | Day 0, Day 14, Day 28
Fasting hematology profile: neutrophil count | Day 0, Day 14, Day 28
Fasting hematology profile: red blood cell count | Day 0, Day 14, Day 28
Fasting hematology profile: hemoglobin | Day 0, Day 14, Day 28
Fasting hematology profile: hematocrit | Day 0, Day 14, Day 28
Fasting hematology profile: platelet count | Day 0, Day 14, Day 28
Fasting blood lipid profile: triglycerides | Day 0, Day 14, Day 28
Fasting blood lipid profile: total cholesterol | Day 0, Day 14, Day 28
Fasting blood lipid profile: LDL-C | Day 0, Day 14, Day 28
Fasting blood lipid profile: non HDL-C | Day 0, Day 14, Day 28
Fasting blood lipid profile: HDL-C | Day 0, Day 14, Day 28
Fasting serum chemistry: chlorides | Day 0, Day 14, Day 28
Estimated glomerular filtration rate | Day 0, Day 14, Day 28
Fasting serum chemistry: direct bilirubin | Day 0, Day 14, Day 28
Fasting hematology profile: mean corpuscular volume | Day 0, Day 14, Day 28
Fasting hematology profile: mean corpuscular hemoglobin | Day 0, Day 14, Day 28
Fasting hematology profile: mean corpuscular hemoglobin concentration | Day 0, Day 14, Day 28
Fasting hematology profile: red cell distribution width | Day 0, Day 14, Day 28
Fasting hematology profile: mean platelet volume | Day 0, Day 14, Day 28
Fasting hematology profile: lymphocyte concentration | Day 0, Day 14, Day 28
Fasting hematology profile: monocyte count | Day 0, Day 14, Day 28
Fasting hematology profile: eosinophil count | Day 0, Day 14, Day 28
Fasting hematology profile: basophil count | Day 0, Day 14, Day 28
Fasting hematology profile: immature granulocytes count | Day 0, Day 14, Day 28
Fasting hematology profile: immature granulocytes (% of WBC) | Day 0, Day 14, Day 28
Fasting hematology profile: neutrophil (% of WBC) | Day 0, Day 14, Day 28
Fasting hematology profile: lymphocyte (% of WBC) | Day 0, Day 14, Day 28
Fasting hematology profile: monocyte (% of WBC) | Day 0, Day 14, Day 28
Fasting hematology profile: eosinophil (% of WBC) | Day 0, Day 14, Day 28
Fasting hematology profile: basophil (% of WBC) | Day 0, Day 14, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Marc Surette, PhD, Principal Investigator — Université de Moncton; Rémi LeBlanc, MD, Principal Investigator — Centre Hospitalier Dr Georges-L.-Dumont
Locations (1):
- Université de Moncton, Moncton, New Brunswick, Canada